CLINICAL TRIAL: NCT03855787
Title: Ureteral Stent Placement After Ureteroscopy for Renal Stones: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Université de Montréal (Other); University of California, Davis (Other); University of California, San Diego (Other); Indiana University (Other); Brigham and Women's Hospital (Other); Penn State Health (Unknown); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Ryan Hsi, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: URSSTONE
Record Dates: First submitted 2019-02-24; First posted 2019-02-27 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi | interventions — Ureteroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ureteral stent group (Active Comparator): A ureteral stent will be placed after ureteroscopy.
  Interventions: Procedure: Ureteroscopy
- No ureteral stent group (Active Comparator): A ureteral stent will not be placed after ureteroscopy.
  Interventions: Procedure: Ureteroscopy

INTERVENTIONS:
Procedure: Ureteroscopy — Ureteroscopy for 1.5cm or less renal stones.
  Other Names: Flexible ureteroscopy

SUMMARY:
The rationale for this study is to determine if there is a difference in complications among patients undergoing ureteroscopy for renal stones who receive a stent compared to not receiving a stent postoperatively.

DETAILED DESCRIPTION:
Kidney stones affect 9% individuals within the United States, and the prevalence is increasing. Over the last few decades, ureteroscopy has become the most commonly performed stone procedure. However the complication rate after ureteroscopy is not insignificant. Reducing morbidity after ureteroscopy would improve patient outcomes and reduce health care utilization.

A major contributor to patient morbidity after ureteroscopy is the ureteral stent, which is placed at the time of surgery and left in place 1-2 weeks after surgery. The rationale for utilizing stents is to prevent urinary obstruction from edema or stone fragments. On the other hand, stents cause hematuria, pain, and lower urinary tract symptoms. Additionally, stent-related symptoms are often misdiagnosed as urinary tract infections leading to unnecessary antibiotic use.

The clinical utility of ureteral stents after ureteroscopy has not been well studied, specifically a stone located in the kidney. Prior studies on stent-less ureteroscopic procedures have focused on treatment of ureteral stones and not stones located in the kidney, have had restrictive inclusion and exclusion criteria, are primarily from single center institutions, and most being performed ~15 years ago. Surgical techniques and device innovations have changed the procedure since that time. To date, there have been only 2 studies that included stone located in the kidney showing no difference in unplanned hospital revisits, however both combined analyses with ureteral stones and selection bias was an issue for both studies. In addition, there is a lack of studies assessing opiate use, impact of quality of life with stent placement, and loss of work related to stent placement

ELIGIBILITY:
Inclusion Criteria:

* nonobstructing renal stone 1.5cm total stone diameter (if multiple stones, then sum of maximum diameters) or less undergoing ureteroscopy

Exclusion Criteria:

* age < 18 years
* pregnancy status
* ureteral stone
* preoperative hydronephrosis
* indwelling nephrostomy tube
* planning bilateral ureteroscopy or subsequent staged ureteroscopy
* solitary kidney or eGFR <60 mL/min (CKD stage 3 or greater)
* variant anatomy including horseshoe kidney, pelvic kidney, prior urinary tract reconstruction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 103 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Total number of complications | 30 days after ureteroscopy
  Total number of complications - Defined as ER visits related to procedure, unanticipated provider visit, and hospitalization

SECONDARY OUTCOMES:
PROMIS (Patient-Reported Outcomes Measurement Information System) form 6a | baseline to 5-10 days after ureteroscopy
  This survey assesses self-reported consequences of pain on relevant aspects of one's life, including engagement with social, cognitive, emotional, physical, and recreational activities. There are 6 questions on the survey. The survey score uses at T-score metric with a mean of 50 and a standard deviation of 10 in a referent population. A higher score denotes greater pain interference in one's life.
WISQOL (Wisconsin Stone Quality of Life Questionnaire) | baseline to 5-10 days after ureteroscopy
  This is a disease specific quality-of-life instrument designed to assess the impact on patients of stones in the urinary tract. The survey is a 28-item instrument with a 5-point LIkert scale for each item. There are a total of 140 points total, and a difference of 10 points can be considered clinically significant.
Cumulative opiate morphine equivalent dosing (MED) | baseline to 5-10 days after ureteroscopy
  This will be the calculated morphine equivalent dosage of all opiate medications that are prescribed after surgery to follow-up at 5-10 days.
% return to work | 5-10 days after ureteroscopy
  This is the number of participants that have returned to work at the time of follow-up at 5-10 days divided by the total participants in the group.
Number of participants with symptomatic urinary tract infection (UTI) | Baseline 5-10 days after ureteroscopy
  This will be defined as a urine culture positivity (50,000 cfu/mL or more) with urinary symptoms.
Number of participants with abnormal imaging findings | 4-8 weeks after ureteroscopy
  Hydronephrosis, hematoma, urinoma on routine postop imaging

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Hsi, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (7):
- United States (6):
  - University of California Los Angeles, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of California San Diego, San Diego, California
  - Indiana University Health Physicians Urology, Indianapolis, Indiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Vanderbilt University Medical Center, Nashville, Tennessee
- University of Montreal, Montreal, Canada

IPD SHARING:
Plan to Share IPD: No